CLINICAL TRIAL: NCT03073746
Title: Accuracy of Differential Diagnosis From Google Health Search and Impact on Clinical Encounters
Brief Title: Google Health Search Trial
Acronym: GHST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Google LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00088552
Record Dates: First submitted 2017-02-16; First posted 2017-03-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diagnoses Disease
Keywords: Google; Knowledge Panels; Health Search; Online; Internet; Smartphone; Tablet; Digital; Mobile; Symptoms; Differential diagnosis; Diagnosis; Anxiety
MeSH Terms: conditions — Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants presenting with new symptoms to either an urgent care center or emergency department will be randomized in a 1:1:1 ratio to one of three groups. 1. Access to Health Search (i.e. Google's new health search platform for mobile devices; Health Knowledge Panels and Symptom Search Tool); 2. Access to Standard Search (i.e. prior version of Google search); 3. Usual Care. Groups 1 and 2 will use a tablet or mobile phone to search while group 3 will not.
Who Masked: Care Provider
Masking Description: Healthcare providers will not have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Search (Experimental): Access to Health Knowledge Panels and Symptom Search Tool.
  Interventions: Other: Health Search
- Standard Search (Experimental): No access to Health Knowledge Panels and Symptom Search Tool, but access to prior version of Google search.
  Interventions: Other: Standard Search
- No Search (No Intervention): No access to Health Knowledge Panels, Symptom Search Tool, prior version of Google search, or mobile device.

INTERVENTIONS:
Other: Health Search
  Arms: Health Search
Other: Standard Search
  Arms: Standard Search

SUMMARY:
There are large differences in knowledge between patients and healthcare providers (i.e. physicians, physician assistants and nurse practitioners), and there is a strong interest on the part of both industry and academia to reduce the gap in knowledge between patients and healthcare providers. Currently, about 1 in 20 searches on Google are health related. Among internet users, 72% reported searching for health information, and among persons who use mobile phones, 31% of cell phone users and 52% of smartphone users have looked up health or medical information. Oftentimes, patients will search on Google or other search engines in order to find health conditions that explain their symptoms prior to visiting their healthcare provider. With the launch of Google's new health search tools for mobile devices (i.e. smartphones, tablets, etc.) it is important to understand how patients use these search platforms and what their effects are on clinical encounters. The main objective of this study is to understand the accuracy of differential diagnoses generated by Google searching; the investigators hypothesize that searching on Google using a tablet or mobile device will be more accurate than not using any search tool, and that the new health search experience will improve accuracy over the standard search platform.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient >= 18 years of age
* Presenting for care at urgent care or emergency department
* In search of a diagnosis to explain a new symptom or group of symptoms

Exclusion Criteria:

* Not literate, defined as lacking the ability to read and write (self-reported)
* Non-English Speaking (self-reported)
* Not mentally competent to provide consent due to inability to understand relevant information due to deficit in intelligence (e.g. mental retardation), memory (e.g., advanced dementia or significant delirium), or attention span (e.g., Attention Deficit Disorder (ADD) or mania) based on prior documentation in medical records or as judged by the researchers)
* Unable to use phone/tablet for any mental or physical impairment (e.g., blind) (self-reported)
* Exacerbation of chronic condition (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of patient's pre-visit differential diagnosis after Google searching on a tablet or mobile phone. | Assessing diagnostic accuracy from baseline to up to one hour post-clinical encounter.
  Proportion of patient's pre-visit differential diagnosis meeting the criteria of "match" with clinician post-visit differential diagnosis (i.e. Two of the three conditions on the clinician's differential diagnosis were more likely to be present in the patient's pre-visit assessment when a tablet or mobile phone was present).

SECONDARY OUTCOMES:
Accuracy of differential diagnosis of Health Search vs. Standard Search | Assessing diagnostic accuracy from baseline to up to one hour post-clinical encounter.
  Proportion of patient's pre-visit differential diagnosis meeting the criteria of "match" with clinician post-visit differential diagnosis comparing Arm 1 (i.e. Health Search) vs. Arm 2 (i.e. Standard Search).

OTHER OUTCOMES:
Changes in anxiety on a visual analog scale | Assessing a change in anxiety from baseline to up to one hour post clinical encounter.
  Comparing changes in anxiety (pre-clinical encounter vs. post-clinical encounter) among treatment arms. (Health Search vs. Standard Search).

CONTACTS AND LOCATIONS:
Overall Officials: Seth S Martin, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Background] "Health Fact Sheet." Pew Research Center, Washington D.C. (December 16, 2013). http://www.pewinternet.org/fact-sheets/health-fact-sheet/.